CLINICAL TRIAL: NCT03132168
Title: Postoperative Delirium in Patients Undergoing Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ahmad Shabsigh, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016H0021
Record Dates: First submitted 2017-04-05; First posted 2017-04-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Post-operative Delirium
Keywords: cystectomy; urology; surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: All consented subjects will be undergoing elective, scheduled surgeries with standardized anesthesia regimen per protocol. Each participant will complete surveys and procedures as outlined per protocol.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects undergoing radical cystectomy (Other): Subjects involved in the study will be evaluated with various non-invasive assessments including the Richmond Agitation-Sedation Scale, pain assessments on a Numeric Rating Scale (NRS-11), and CAM-ICU scale. Blood draws will also take place in order to perform microRNA testing in all subjects participating in the trial. Standardized anesthetic care as described by the approved protocol will be followed for each subject included in this trial.
  Interventions: Behavioral: Assessments; Procedure: Blood Draw; Other: Standardized Anesthetic Care

INTERVENTIONS:
Behavioral: Assessments — These cognitive assessments will be utilized during the study to evaluate cognitive levels comparing prior to surgery and post-operatively in order to determine if the subject is delirious. BIS monitoring will be utilized for all subjects.
  Other Names: SAGE scale, Memorial Delirium Assessment Scale
Procedure: Blood Draw — Subjects will have blood draws at surgical preadmission visit, Day 1, Day 2, and Day 3 post surgery only; one tube containing approximately one teaspoon (5 mL) of blood will be drawn at each visit.
Other: Standardized Anesthetic Care — Standardized anesthetic care will be provided as described by the protocol for each subject consented for this trial.
  Other Names: Anesthetic Regimen

SUMMARY:
In this study, post-operative delirium will be measured in patients undergoing surgery for bladder resection, and associated microRNA biomarkers will be evaluated in patients considered delirious and non-delirious after surgery.

DETAILED DESCRIPTION:
With voluntary participation, this study requires participants to complete a self-administered cognitive evaluation (SAGE) before surgery to assess baseline cognitive impairment and early dementia; vital signs will be documented prior to surgery. During surgery, participants will receive a standardized general anesthesia regimen as described in the protocol. Several parameters will be measured during surgery, including bispectral monitoring to measure processed EEG. After surgery, fitness for cognitive evaluation will be determined by the Richmond Agitation-Sedation Scale (RASS) scale, and then emergence delirium will be assessed using the CAM-ICU scale. Fitness for discharge from PACU will be determined by an Aldrete score of 9 or more. Postoperative pain will be assessed using the 11-point Numeric Rating Scale (NRS-11). Postoperative nausea and vomiting (PONV) level will also be documented. Postoperative Delirium (POD) assessment will be achieved by administering the memorial delirium assessment scale (MDAS) twice a day starting on day 1 through day 3 postoperatively. Pain NRS-11 score and PONV levels will also be documented at each visit. For microRNA testing, blood probes will be collected in 5mL purple top tube at surgical preadmission and post-surgery days one, two and three. Risks associated with participating in this study include normal risk associated with having surgery and general anesthesia; no greater than minimal risk is associated with blood collection. For the participant, there are no immediate anticipated benefits for participating in this study. The importance of the knowledge that is expected to result includes lower post-operative complications as a result of post-operative delirium, faster recovery, and shorter hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age and older
* ASA II or III
* Capable of and willing to consent
* Participants literate in English language

Exclusion Criteria:

* ASA IV or V
* Patients with severe visual or auditory impairment
* Inability to read and/or write in English
* Presence of a clinically diagnosed major psychiatric condition such as bipolar disorder, uncontrolled major depression, schizophrenia
* Dementia of Alzheimer's type
* Parkinson's disease
* Multiple Sclerosis (MS)
* Vascular dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Post-operative delirium | up to 3 days post-operatively
  Evaluate the incidence of and risk factors for POD in patients undergoing radical cystectomy utilizing the Memorial Delirium Assessment Scale.

SECONDARY OUTCOMES:
microRNA expression | up to 3 days post-operatively
  A secondary aim of the study is to obtain estimates and variances of the difference in microRNA expression between 2 groups: delirious patients and non-delirious patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Shabsigh, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No